CLINICAL TRIAL: NCT00035971
Title: EVA: Evista Alendronate Comparison
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 5548; H3S-US-GGKO
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: raloxifene HCI and alendronate Na

SUMMARY:
The purpose of this study is to determine how treatment with raloxifene compares to treatment with alendronate in postmenopausal women with osteoporosis on the chance of experiencing fractures

ELIGIBILITY:
Inclusion Criteria

* 50-80 years of age, inclusive
* 2 years since last menses
* Dx femoral neck osteoporosis
* No vertebral fractures

Exclusion Criteria

* Poor candidate for study drugs
* Hx of diseases affecting bone metabolism
* Hx of breast/estrogen-dependent cancer
* Current use of osteoporosis drug therapy
* Hx/high risk of VTE

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (86):
- United States (73):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Anniston, Alabama
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Loma Linda, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Oakland, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Walnut Creek, California
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Lakewood, Colorado
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Maitland, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Fayetteville, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Gainesville, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Riverdale, Georgia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Honolulu, Hawaii
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Idaho Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Morton Grove, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Evansville, Indiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Des Moines, Iowa
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Frederick, Maryland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Hagerstown, Maryland
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Springfield, Missouri
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Lebanon, New Hampshire
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Passaic, New Jersey
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Albany, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Greensboro, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Morehead City, North Carolina
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY(1-877-285-4559) or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Johnston, Rhode Island
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559 or speak with your personal physician., Temple, Texas
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Charlottesville, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Newport News, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Spokane, Washington
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support Center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Madison, Wisconsin
- Canada (13):
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Moncton, New Brunswick
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Burlington, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Kitchener, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Ottawa, Ontario
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Trois-Rivières, Quebec
  - For additional information regarding investigative sites for this trial, contact the Clinical Trials Support center at 1-877-CTLILLY (1-877-285-4559) or speak with your personal physician., Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Recker RR, Kendler D, Recknor CP, Rooney TW, Lewiecki EM, Utian WH, Cauley JA, Lorraine J, Qu Y, Kulkarni PM, Gaich CL, Wong M, Plouffe L Jr, Stock JL. Comparative effects of raloxifene and alendronate on fracture outcomes in postmenopausal women with low bone mass. Bone. 2007 Apr;40(4):843-51. doi: 10.1016/j.bone.2006.11.001. Epub 2006 Dec 19. PMID 17182297